CLINICAL TRIAL: NCT02770508
Title: A Phase 4, Randomized, Open Label, Controlled Study of Boosted Darunavir and Lamivudine Versus Boosted Darunavir and Emtricitabine/Tenofovir or Lamivudine/Tenofovir in Naïve HIV-1 Infected Subjects
Brief Title: Darunavir/Ritonavir + Lamivudine Versus Darunavir/Ritonavir +Emtricitabine/Tenofovir in Naïve HIV-1 Infected Subjects
Acronym: ANDES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Huésped (Other)
Collaborators: Ministry of Science and Technology,Argentine (Unknown); National AIDS and STD programme,Argentine (Unknown); Richmond Laboratories (Unknown)
Responsible Party: Principal Investigator, Pedro Cahn, PhD, MD, Fundación Huésped
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FH-15
Record Dates: First submitted 2015-11-16; First posted 2016-05-12 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: HIV-1 Infection
Keywords: antiretroviral naive; dual therapy
MeSH Terms: interventions — Darunavir; Ritonavir; Lamivudine; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Darunavir/ritonavir plus lamivudine (Experimental): Darunavir/ritonavir 800/100 mg, 1 coformulated tablet QD and lamivudine 300 mg, 1 tablet QD
  Interventions: Drug: darunavir/ritonavir; Drug: Lamivudine
- Darunavir/ritonavir plus emtricitabine/tenofovir(FTC/TFD) (Active Comparator): Darunavir/ritonavir 800/100 mg1 coformulated tablet QD (FDC) plus FTC/TDF 200/300 mg, 1 coformulated tablet QD
  Interventions: Drug: darunavir/ritonavir; Drug: emtricitabine-tenofovir(FTC/TDF)

INTERVENTIONS:
Drug: darunavir/ritonavir
  Other Names: Virontar R
Drug: Lamivudine
  Other Names: 3TC
  Arms: Darunavir/ritonavir plus lamivudine
Drug: emtricitabine-tenofovir(FTC/TDF)
  Other Names: TRUVADA
  Arms: Darunavir/ritonavir plus emtricitabine/tenofovir(FTC/TFD)

SUMMARY:
The purpose of this study is to compare the safety and efficacy of a combination of a QD regimen consisting on ritonavir boosted darunavir (FDC) and lamivudine versus ritonavir boosted darunavir (FDC) plus co-formulated tenofovir and emtricitabine or co-formulated tenofovir/lamivudine in naïve HIV-1 infected patients. Subjects will be ARV-naïve HIV-1-infected patients eligible to start ARV therapy according to current guidelines.Subjects will be adults ≥ 18 years of age who meet all of the inclusion criteria and none of the exclusion criteria.

DETAILED DESCRIPTION:
Key Inclusion Criteria

1. Documented HIV RNA >1000 copies/ml
2. Subject naïve to ARV. .
3. Subject has indication to receive an antiretroviral regimen, based on local guidelines.
4. Able to provide informed consent and agree to use a highly effective non-hormonal method of contraception

Key Exclusion Criteria

1. Evidence of resistance to Darunavir and/or FTC or 3TC or TDF based on the resistance test
2. Patient with chronic hepatitis B
3. Subject has a currently active AIDS defining illness (Category C conditions according to the CDC Classification System
4. Required use of disallowed concomitant therapies
5. Subject with the grade 3 or 4 laboratory abnormalities as defined by DAIDS grading table

Primary Objective

• Proportion of patients with HIV-1 RNA levels of less than 50 copies/mL at week 48 (ITT analysis, Snapshot analysis)

ELIGIBILITY:
Inclusion criteria :

1. > 18 years of age.
2. Patient with documented HIV-1 infection defined as a positive ELISA plus a confirmatory Western Blot; or alternatively, a plasma HIV-1 RNA ≥1,000 copies/mL ever documented.
3. Subject has voluntarily signed and dated an informed consent form, approved by an Institutional Review Board (IRB) / Independent Ethics Committee (IEC), after the nature of the study has been explained and the subject has had the opportunity to ask questions. The informed consent must be signed before any study-specific procedures are performed.
4. Subject agrees not to take any medication during the study, including over the counter medicines or herbal preparations, without the approval of the trial physician.
5. Documented HIV-1 RNA >1,000 copies/mL
6. Subject naïve to ARV. (Patients who had received ARV ≤ 48 hours are allowed). Subject has indication to receive an antiretroviral regimen.
7. Subjects can comply with protocol requirements.
8. Subject's general medical condition, in the investigator's opinion, does not interfere with assessments and completion of the trial.
9. If patient is a female she must not be breastfeeding or pregnant. She must be either postmenopausal for at least one year, surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy), or she must:

   * use 2 different methods of birth control including, at least, one barrier method, and are acceptable to both the subject and investigator, and
   * has a urine pregnancy test performed at the Screening Visit and on Baseline. Results of both tests must be negative.
   * continue using 2 different methods of birth control including, at least, one barrier method for at least 30 days after the end of the treatment period
10. For male patients, must comply with the use of a barrier birth control method during the Study and 60 days beyond the Study completion

Exclusion criteria :

1. Evidence of resistance to or 3TC or DRV/r, TDF, FTC o 3TC based in the results of the resistance testing done in the screening visit, such resistance being considered in accordance with IAS-USA panel, version dated March 2013.

   Any of the following mutations will be considered resistance to DRV/r :
   * I47V, I50V, I54M/L, L76V, I84V or, 3 or more minor mutations : V11I, V32I, L33F, T74P, L89V.
   * Any of the following mutations will be considered resistance to 3TC or FTC : M184V/I and /or K65R and / or Q151M.
   * Any of the following mutations will be considered resistance to TDF: K65R, K70E, double insertion 69 or 3 TAMS including M41L or L210W.
2. Prior HIV-2 documented infection.
3. The use of disallowed concomitant therapy (see Appendix C).
4. Active Hepatitis B infection (at any stage).
5. The patient was diagnosed with acute active hepatitis by any cause, or chronic hepatitis C WITH levels of aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 5 higher than the upper limit of normal (ULN) AND/OR may require one-year treatment.
6. Any clinical significant active disease (for instance, tuberculosis, heart failure, pancreatitis) or any medical history or physical examination findings that, according to the investigator's opinion, may risk the patient's safety, the results of the study or adherence to the rules of the protocol.
7. The patient has an active AIDS-associated opportunistic disease (Category C according to the CDC classification system for HIV infection as of 1993) within 30 days after the screening. Stabilized patients under treatment for AIDS-associated opportunistic disease may be included in the study.
8. Life expectancy < 1 year according to the investigator
9. Laboratory tests performed during the screening visit show any of the following alterations:

   * Hemoglobin <8.0 gm/dL
   * Absolute neutrophil count (ANC) < 750 cells/µL
   * Platelet Count < 50,000 cells/mm3
10. The use of any study agent within 30 days as from the screening.
11. Use of immunosuppressive drugs, cytokines inhibitors or other cytokines over the prior year.
12. Any other condition (including, without limitation, the use of alcohol or drugs) that in the investigator's opinion may compromise the safety of the patient or his/her adherence to the protocol
13. Patients who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2015-11; Primary Completion 2017-07 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with HIV-1 RNA levels of less than 50 copies/mL at week 48 | 48 weeks
  The percentage of participants with Plasma Human Immunodeficiency Virus-1 (HIV-1) <50 c/mL at Week 48 will be assessed using Missing, Switch or Discontinuation = Failure (MSDF), as codified by the Food and Drug Administration (FDA) "snapshot" algorithm. This algorithm treated all participants without HIV-1 RNA data at Week 48 as nonresponders, Otherwise, virologic success or failure will be determined by the last available HIV-1 RNA assessment while the participant was on-treatment in the snapshot window (Week 48 +/- 6 weeks).

SECONDARY OUTCOMES:
Percentage of patients with HIV-1 RNA <400 copies/mL at week 24 | 24 weeks
  The percentage of participants with Plasma Human Immunodeficiency Virus-1 (HIV-1) <400 c/mL at Week 24 will be assessed using Missing, Switch or Discontinuation = Failure (MSDF), as codified by the Food and Drug Administration (FDA) "snapshot" algorithm.
Number and type of resistance mutations in case of virologic failure | from week 24 to week 48
  An genotiping test will be made at time to virological failure to detect mutation across reverse transcriptase (RT), and Protease (PRO). Protocol defined virological failure was defined as confirmed plasma HIV-1 RNA levels >=400 copies/mL on or after Week 24 or confirmed plasma HIV-1 RNA levels >=50 copies/mL at week 48
CD4+ lymphocyte count and change between baseline (defined as the average between screening and baseline visit values) and weeks 24 and 48 | week 24 and 48
  Change from Baseline in CD4+ cell counts will be assessed at Weeks 24 and 48.
Frequency, type and severity of adverse events and laboratory abnormalities. | week 24 and 48
  Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment
Clinical disease progression (CDP) | week 24 and 48
  Clinical disease progression (CDP) was assessed according to the Centers for Disease Control and Prevention (CDC) HIV-1 classification system. Category (CAT) A: one or more of the following conditions (CON), without any CON listed in Categories B and C: asymptomatic HIV infection, persistent generalized lymphadenopathy, acute (primary) HIV infection with accompanying illness or history of acute HIV infection. CAT B: symptomatic CON that are attributed to HIV infection or are indicative of a defect in cell-mediated immunity; or that are considered by physicians to have a clinical course or to require management that is complicated by HIV infection; and not included among CON listed in clinical CAT C. CAT C: the clinical CON listed in the AIDS surveillance case definition. Indicators of CDP were defined as: CDC CAT A at Baseline (BS) to a CDC CAT C event (EV); CDC CAT B at BS to a CDC CAT C EV; CDC CAT C at BS to a new CDC CAT C EV; or CDC CAT A, B, or C at BS to death.
Changes in quality of life | baseline, week 24 and week 48
  The evaluation of quality of life will be done through two validated instruments: the Medical Outcomes Study HIV Health Survey ( MOS - HIV) and EuroQol 5D (EQ - 5D ) . Both instruments will be administered to patients at baseline , week 24 and week 48 .

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Cahn, PhD, MD, Principal Investigator — Fundacion Huesped
Locations (5):
- Argentina (5):
  - Consultorio Infectológico Dr. Pryluka, CABA, Buenos Aires
  - Hospital Cosme Argerich, CABA, Buenos Aires
  - Hospital Italiano, CABA, Buenos Aires
  - Fundacion huesped, CABA, Buenos Aires
  - Centro de Estudios Infectologicos SA (CTD Stamboulian), CABA, Buenos Aires

IPD SHARING:
Plan to Share IPD: Yes
To publish week 48 study

REFERENCES:
- [Derived] Figueroa MI, Sued O, Cecchini D, Sanchez M, Rolon MJ, Lopardo G, Ceschel M, Mernies G, De Stefano M, Patterson P, Gun A, Fink V, Ortiz Z, Cahn P; ANDES Study Group. Dual therapy based on co-formulated darunavir/ritonavir plus lamivudine for initial therapy of HIV infection: The ANDES randomized controlled trial. Int J Antimicrob Agents. 2024 Oct;64(4):107301. doi: 10.1016/j.ijantimicag.2024.107301. Epub 2024 Aug 14. PMID 39151647